CLINICAL TRIAL: NCT04806243
Title: A Phase II, Second-line, Single-arm Clinical Trial of Carelizumab Combined With Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Carelizumab Combined With Regorafenib in the Treatment of HCC（CARE-2020）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-010
Record Dates: First submitted 2021-03-04; First posted 2021-03-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carelizumab Combined With Regorafenib arm (Experimental)
  Interventions: Drug: Regorafenib Pill&Camrelizumab

INTERVENTIONS:
Drug: Regorafenib Pill&Camrelizumab — Regorafenib，80 mg，QD，Q3w Camrelizumab，200 mg，IV，Q3w

SUMMARY:
To investigate the efficacy and safety of carelizumab combined with regorafenib in second-line treatment for patients with primary hepatocellular carcinoma.

DETAILED DESCRIPTION:
Currently, there is little experience in the application of targeted drugs combined with immunotherapy. Through this study, we hope to explore the optimal population for the use of carelizumab combined with regorafenib in the second-line treatment of hepatocellular carcinoma (HCC), as well as the efficacy and safety.

This research is a single-center trials phase II second-line, single arm, explore the clinical outcome of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Not convenient to disclose

Exclusion Criteria:

* Not convenient to disclose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
os（overall survival） | 21 days
  overall survival

SECONDARY OUTCOMES:
PFS（progression-free survival） | 21 days
  progression-free survival
TTP（Time-To-Progression） | 21 days
  Time-To-Progression
ORR（Overall Response Rate） | 21 days
  Overall Response Rate
DCR（disease control rate） | 21 days
  disease control rate
DoR | 21 days
  Duration of Response

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No